CLINICAL TRIAL: NCT05007925
Title: Prospective, Multi-center, Single-arm Study of the Shockwave Medical Peripheral Intravascular Lithotripsy (IVL) System for Treatment of Calcified Peripheral Arterial Disease (PAD) in Below-the-Knee (BTK) Arteries
Brief Title: Disrupt PAD BTK II Study With the Shockwave Peripheral IVL System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 65007
Record Dates: First submitted 2021-08-09; First posted 2021-08-17 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single-arm (Experimental)
  Interventions: Device: Intravascular Lithotripsy

INTERVENTIONS:
Device: Intravascular Lithotripsy — Localized peripheral intravascular lithotripsy

SUMMARY:
To assess the continued safety, effectiveness, and optimal clinical use of the Shockwave Medical Peripheral IVL System for the treatment of calcified, stenotic BTK arteries.

Post-market, prospective , multi-center, single-arm study.

ELIGIBILITY:
Inclusion Criteria:

- General Inclusion Criteria

1. Age of subject is ≥ 18.
2. Subject is able and willing to comply with all assessments in the study.
3. Subject or subject's legal representative has been informed of the nature of the study, agrees to participate, and has signed the approved consent form.
4. Critical limb ischemia (CLI) in the target limb from the distal segment (P3) of the popliteal artery to the ankle joint prior to the study procedure with Rutherford Category 4-5; or Rutherford 3 in the target limb from the distal segment (P3) of the popliteal artery to the ankle joint prior to the study procedure.
5. Estimated life expectancy >1 year.

   * Angiographic Inclusion Criteria
6. Up to 2 below-the-knee target lesion(s) in native vessels in one or both limbs.
7. Target lesion reference vessel diameter (RVD) between 2.0 mm and 4.0 mm by investigator visual estimate.
8. Target lesion with ≥70% stenosis by investigator visual estimate.
9. Target lesion length is ≤200 mm by investigator visual estimate. Target lesion can be all or part of the 200 mm treated zone.
10. Distal reconstitution of at least one pedal vessel (<50% stenosis) (desert foot excluded).
11. Evidence of at least moderate calcification at the target lesion site by angiography/IVUS OR non-dilatable lesion indicating presence of calcium. Must meet one of the following:

    1. Angiography requires fluoroscopic evidence of calcification on parallel sides of the vessel and extending > 50% the length of the lesion.
    2. IVUS requires presence of ≥270 degrees of calcium over the course of at least 10mm.
    3. Non-dilatable lesion requires attempted treatment with PTA during the index procedure with residual stenosis > 50% and no serious angiographic complications.

Exclusion Criteria:

- General Exclusion Criteria

1. Rutherford Category 0, 1, 2 or 6 (target limb).
2. Osteomyelitis or deep soft tissue infection extending proximal from the metatarsals that cannot be treated with an individual toe ray amputation or transmetatarsal amputation (TMA) .
3. History of endovascular or surgical procedure on the target limb within the last 30 days, or planned within 30 days of the index procedure.
4. Subject in whom antiplatelet or anticoagulant therapy is contraindicated.
5. Subject has known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
6. Subject has known allergy to urethane, nylon, or silicone.
7. Myocardial infarction within 30 days prior to enrollment.
8. History of stroke within 60 days prior to enrollment.
9. Subject has acute or chronic renal disease with eGFR <30 ml/min/1.73 m2 (using CKD-EPI formula), unless on renal replacement therapy.
10. Subject is pregnant or nursing.
11. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.
12. Subject has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.
13. Covid-19 diagnosis within 90 days.
14. The planned use of cutting/scoring balloons, re-entry or atherectomy devices in target lesions during the index procedure.
15. Planned major amputation (of either leg).
16. Acute limb ischemia.
17. Occlusion of all the inframalleolar outflow arteries/vessels (i.e., desert foot).
18. Subject has an anticipated life span of less than one (1) year.
19. Subject already enrolled into this study.

    * Angiographic Exclusion Criteria
20. Failure to treat clinically significant inflow lesions in the ipsilateral iliac, femoral, or popliteal arteries with ≤30% residual stenosis, and no serious angiographic complications (e.g., embolism).
21. Failure to successfully treat significant non-target infra-popliteal lesions prior to treatment of target lesion(s). Successful treatment is defined as obtaining ≤50% residual stenosis with no serious angiographic complications (e.g., embolism ).
22. Failed PTA in target lesion during index procedure with angiographic evidence of serious angiographic complications .
23. Target lesion includes in-stent restenosis.
24. Evidence of aneurysm or thrombus in target vessel.
25. No calcium or mild calcium in the target lesion.
26. Target lesion within native or synthetic vessel grafts.
27. Failure to successfully cross the guidewire across the target lesion; successful crossing defined as tip of the guidewire distal to the target lesion in the absence of flow limiting dissections or perforations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2026-04-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (39):
  - UCSF Fresno, Fresno, California
  - Scripps Memorial Hospital, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford Hospital, Palo Alto, California
  - UC Davis Health, Sacramento, California
  - St. Helena Hospital, St. Helena, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Medstar Montgomery Medical Center, Olney, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Southcoast Hospitals Group, New Bedford, Massachusetts
  - McLaren Bay Heart and Vascular, Bay City, Michigan
  - McLaren Greater Lansing, Lansing, Michigan
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - NYU Langone Medical Center, New York, New York
  - Mt. Sinai Hospital, New York, New York
  - Columbia University Irving Medical Center/NYPH, New York, New York
  - Charlotte Radiology, Charlotte, North Carolina
  - North Carolina Heart & Vascular, Raleigh, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Ascension St Johns Heart & Vascular Center, Bartlesville, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Harrisburg, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Wellmont Cardiology Services dba CVA Heart Institute, Kingsport, Tennessee
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Texas Health Presbyterian Hospital, Dallas, Texas
  - Baylor Scott & White - The Heart Hospital Baylor, Plano, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - VA Puget Sound Health Care Systems - Seattle, Seattle, Washington
- Germany (4):
  - Karolinen-Hospital Hüsten, Arnsberg
  - Universitäts-Herzzentrum Freiburg & Bad Krozingen, Bad Krozingen
  - Universitätsklinikum der Ruhr-Universitaet Bochum, Bad Oeynhausen
  - Universitätsklinikum Leipzig AoR, Leipzig

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Lesions
Groups:
- Disrupt PAD BTK II: Disrupt PAD BTK II: Prospective, Multi-center, Single-arm Study of the Shockwave Medical Peripheral Intravascular Lithotripsy (IVL) System for Treatment of Calcified Peripheral Arterial Disease (PAD) in Below-the-Knee (BTK) Arteries
Period: Overall Study
Arm/Group | Disrupt PAD BTK II
Started | 250; 305 Lesions
Completed | 242; 303 Lesions
Not Completed | 8; 2 Lesions

BASELINE CHARACTERISTICS:
Arm/Group | Disrupt PAD BTK II
Number analyzed (Participants) | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 63
  >=65 years | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 182
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 45
  White | 181
  Unknown or Not Reported | 14
  Other | 4
Region of Enrollment [Number; unit: participants]
  United States | 239
  Germany | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedure Success
Description: Procedure Success defined as ≤50% residual stenosis for all treated target lesions without serious angiographic complications (flow-limiting dissection, perforation, distal embolization, or acute vessel closure) as assessed by the angiographic core lab at the final timepoint.
Time Frame: 30 days
Population: The final procedure success at the subject level was 97.9% (232/237). There were five subjects (one subject had both angiographic complications and ≤ 50% residual stenosis) that did not have procedure success. There were three subjects with serious angiographic complications: two subjects had a grade I perforation and one subject had both an abrupt closure and grade F dissection.
Measure: Count of Participants; unit: Participants
Groups:
- Shockwave Medical M5, M5+, S4 Peripheral Intravascular Lithotripsy System: The Shockwave Medical IVL System is intended for lithotripsy-enhanced balloon dilatation of lesions, including calcified lesions, in the peripheral vasculature, including the iliac, femoral, ilio-femoral, popliteal, infra-popliteal, and renal arteries. Not for use in the coronary or cerebral vasculature.
Arm/Group | Shockwave Medical M5, M5+, S4 Peripheral Intravascular Lithotripsy System
Number analyzed (Participants) | 237
Participants | 232

2. Primary Outcome: Number of Participants With Major Adverse Limb Events (MALE) + Post-Operative Death (POD)
Description: Major Adverse Limb Events (MALE) + Post-Operative Death (POD) at 30 days defined as a composite of:
  * all-cause death
  * above-ankle amputation of the index limb
  * major reintervention (new bypass graft, jump/interposition graft revision, or thrombectomy/thrombolysis) of the index limb involving a BTK artery
Time Frame: 30 days
Population: There were two (0.8%, 2/242) MALE events at 30 days that were adjudicated as above-ankle amputations of the index limb. Both major amputations were CEC adjudicated as unplanned amputations unrelated to the study procedure and IVL device. There were no deaths or major reinterventions within 30 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5, M5+, S4 Peripheral Intravascular Lithotripsy System
Number analyzed (Participants) | 242
Participants | 2

3. Primary Outcome: Subjects Without Serious Angiographic Complications
Description: Subject Success defined as final residual stenosis ≤ 50% in the target lesion without serious angiographic complications as assessed by the angiographic core lab. Serious angiographic complications include (flow-limiting dissection, perforation, distal embolization, or acute vessel closure) as assessed by the angiographic core lab
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5, M5+, S4 Peripheral Intravascular Lithotripsy System
Number analyzed (Participants) | 237
Participants | 234

4. Secondary Outcome: Number of Lesions With Technical Success
Description: Lesion Success defined as final residual stenosis ≤50% in the target lesion without serious angiographic complications as assessed by the angiographic core lab
Time Frame: 30 days
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Shockwave Medical M5, M5+, S4 Peripheral Intravascular Lithotripsy System
Number analyzed (Participants) | 237
Number analyzed (Lesions) | 290
Lesions
  Lesion Success | 285
  Freedom From Any Serious Angiographic Complications | 287
  Residual Stenosis ≤ 50% | 287

5. Secondary Outcome: Number of Patients With Primary Patency
Description: Primary Patency at 6 and 12 months defined as the absence of both total occlusion (100% diameter stenosis by DUS) in all of the target lesions in a flow pathway, as well as a Clinically-Driven Target Lesion Revascularization (CD-TLR)
Time Frame: 6 and 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Number of Participants Free From Clinically-driven Target Lesion Revascularization (CD-TLR)
Description: Clinically-driven target lesion revascularization (CD-TLR) defined as a composite of:
  * CD-TLR
  * Major target limb amputation
Time Frame: 30 days
Population: The freedom from CD-TLR endpoint at 30 days post-procedure was 99.6% (242/243).
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5, M5+, S4 Peripheral Intravascular Lithotripsy System
Number analyzed (Participants) | 243
Participants | 242

7. Secondary Outcome: Number of Participants With Major Adverse Events (MAE)
Description: Major Adverse Events (MAE) at 30 days defined as a composite of:
  * Need for emergency surgical revascularization of target limb
  * Unplanned target limb major amputation (above the ankle)
  * Symptomatic thrombus or distal emboli that require surgical, mechanical, or pharmacologic means to improve flow, and extend hospitalization
  * Perforations that require an intervention, including bail-out stenting
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5, M5+, S4 Peripheral Intravascular Lithotripsy System
Number analyzed (Participants) | 242
Participants | 5

8. Secondary Outcome: VascuQoL Reported as Change From Baseline
Description: The VascuQoL-6 is a short, disease-specific questionnaire used to measure health-related quality of life (HRQoL) in patients with peripheral arterial disease (PAD), specifically those with intermittent claudication and critical limb ischemia.
Time Frame: 30 days, 6, 12 & 24 months
Reporting Status: Not Posted

9. Secondary Outcome: Ankle-brachial Index (ABI) Reported as Change From Baseline
Description: The ABI is the ratio of systolic blood pressure measured at the ankle to systolic blood pressure measured at the brachial artery. Ideally, this ratio should be 1.0, but is often less in a subject with peripheral arterial disease.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Shockwave Medical M5, M5+, S4 Peripheral Intravascular Lithotripsy System
Number analyzed (Participants) | 158
ratio | 0.2 (0.3)

10. Secondary Outcome: Rutherford Category Reported as Change From Baseline
Description: The Rutherford classification is a system used to categorize the severity of peripheral artery disease (PAD), specifically chronic limb-threatening ischemia (CLTI), based on symptoms and tissue loss. The classification ranges are from Class 0 where no symptoms of PAD are present and the patient has no claudication or tissue loss to Class 6 where patients have extensive tissue loss, including gangrene, that extends above the transmetatarsal level (the area above the bones of the foot). A higher score on the Rutherford Classification Scale is indicative of a worse outcome.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5, M5+, S4 Peripheral Intravascular Lithotripsy System
Number analyzed (Participants) | 227
Participants
  1-Mild Claudication | 21
  2-Moderate Claudication | 14
  3-Severe Claudication | 11
  4-Ischemic Rest Pain | 10
  5- Minor Tissue Loss | 102
  6-Ulceration Or Gangrene | 1
  0-Asymptomatic | 68

11. Secondary Outcome: Toe-brachial Index (TBI) Reported as Change From Baseline
Description: The TBI is the ratio of systolic blood pressure measured at the toe to systolic blood pressure at the brachial artery. Ideally, this ratio should be 1.0, but is often less in a subject with peripheral arterial disease.
Time Frame: 30 Days
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Shockwave Medical M5, M5+, S4 Peripheral Intravascular Lithotripsy System
Number analyzed (Participants) | 9
ratio | 0.2 (0.2)

12. Secondary Outcome: Number of Participants Free From Major Target Limb Amputation
Time Frame: 30 Days
Population: Freedom from amputation at 30 days was assessed in 242 subjects with two subjects experiencing a major target limb amputation within 30 days of index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical M5, M5+, S4 Peripheral Intravascular Lithotripsy System
Number analyzed (Participants) | 242
Participants | 240

ADVERSE EVENTS:
Time Frame: This accounting is for all study events through the 30-day time frame.
Arm/Group | Disrupt PAD BTK II
All-Cause Mortality (participants affected / at risk) | 1/250
Serious Adverse Events (participants affected / at risk) | 67/250
Other Adverse Events (participants affected / at risk) | 131/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Disrupt PAD BTK II (N=250)
Anaemia (Blood and lymphatic system disorders) | 4
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 3
Cardio-respiratory arrest (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haemoperitoneum (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Impaired healing (General disorders) | 7
Ulcer (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Diabetic foot infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 6
Localised infection (Infections and infestations) | 2
Necrotising fasciitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 8
Osteomyelitis chronic (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Septic shock (Infections and infestations) | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 1
Elastic vessel recoil complication (Injury, poisoning and procedural complications) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 4
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1
Vascular access site complication (Injury, poisoning and procedural complications) | 1
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 13
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Malnutrition (Metabolism and nutrition disorders) | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Toe amputation (Surgical and medical procedures) | 1
Dry gangrene (Vascular disorders) | 3
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Intermittent claudication (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 6
Peripheral artery stenosis (Vascular disorders) | 1
Peripheral embolism (Vascular disorders) | 1
Peripheral ischemia (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Disrupt PAD BTK II (N=250)
Anaemia (Blood and lymphatic system disorders) | 4
Cardiac failure congestive (Cardiac disorders) | 3
Impaired healing (General disorders) | 7
Peripheral swelling (General disorders) | 4
COVID-19 (Infections and infestations) | 3
Gangrene (Infections and infestations) | 7
Localised infection (Infections and infestations) | 3
Osteomyelitis (Infections and infestations) | 8
Pneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 6
Limb injury (Injury, poisoning and procedural complications) | 10
Vascular procedure complication (Injury, poisoning and procedural complications) | 59
Hypoglycaemia (Metabolism and nutrition disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Dry gangrene (Vascular disorders) | 3
Haematoma (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT05007925/Prot_SAP_000.pdf